CLINICAL TRIAL: NCT06987214
Title: REGEND001 Autologous Basal Layer Stem Cell Transplantation for Bronchiectasis: A Translational Application Study
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Jieming QU, Professor, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20250514
Record Dates: First submitted 2025-05-14; First posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Bronchiectasis Adult

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bronchiectasis patients (Experimental)
  Interventions: Biological: REGEND001 Autologous Basal Layer Stem Cell Suspension

INTERVENTIONS:
Biological: REGEND001 Autologous Basal Layer Stem Cell Suspension — REGEND001 Autologous Basal Layer Stem Cell Suspension is an innovative cell therapy product designed for chronic structural lung diseases, such as bronchiectasis. This treatment involves harvesting regenerative stem cells (expressing KRT5/P63 markers) from the patient's own bronchial basal layer via fiberoptic bronchoscopy. After isolation, purification, and ex vivo expansion, the cells are administered as a suspension through bronchoscopic infusion into damaged lung segments.

SUMMARY:
This clinical trial aims to evaluate the safety and efficacy of REGEND001, an autologous basal layer stem cell transplantation therapy, in patients with chronic structural lung disease (bronchiectasis). The treatment involves harvesting bronchial basal layer stem cells from the patient, expanding them ex vivo, and reintroducing them via bronchoscopic infusion to repair damaged lung tissue.

ELIGIBILITY:
Inclusion Criteria:

1. Age 25-80 years.
2. Confirmed diagnosis of bronchiectasis.
3. FEV1 ≥35% predicted; DLCO ≥30% and <80% predicted.

Exclusion Criteria:

1. Pregnancy, lactation, or plans for pregnancy within 1 year.
2. Active malignancy or history of malignancy.
3. Positive serology for HIV, HBV, HCV, or syphilis.

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-06-30 (Estimated); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Change in DLCO from baseline. | Baseline, 4 weeks post treatment, 24 weeks post treatment
  The diffusing capacity of the lungs for carbon monoxide (DLCO) is a measurement of the gas transfer capacity of lung.

SECONDARY OUTCOMES:
Change in FEV1 from baseline | Baseline, 4 weeks post treatment, 24 weeks post treatment
  The forced expiratory volume in 1s (FEV1) is a measurement of the airflow capacity.
Incidence of adverse events and serious adverse events. | Through study completion, an average of 6 months
Change in HRCT lung imaging scores | Baseline, 4 weeks post treatment, 24 weeks post treatment
  HRCT, high-resolution computed tomography.
Quality of life (QoL) assessment via validated questionnaires | Baseline, 4 weeks post treatment, 24 weeks post treatment
  Score range: 0 to 100. Higher scores indicate a worse outcome.

IPD SHARING:
Plan to Share IPD: No